CLINICAL TRIAL: NCT04859556
Title: Performance, Safety and Efficiency Comparison Between 10,000 and 5,000 Cuts Per Minute Vitrectomy Using a 25G Cutter - A Prospective Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10K
Record Dates: First submitted 2021-04-20; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Vitreous Hemorrhage; Macula Hole; Epiretinal Membrane; Retinal Detachment
MeSH Terms: conditions — Vitreous Hemorrhage; Retinal Perforations; Epiretinal Membrane; Retinal Detachment

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Patients and Care provider are not able to differentiate the two different cutters since the port size are the exact same for both.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 10k 25G cutter (Experimental): New cutter, with a 10,000 cut per minute blade
  Interventions: Device: Alcon 25Gauge, 10,000 cuts per minute Ultravit cutter
- 5k 25G cutter (Active Comparator): Traditional cutter, with a 5,000 cut per minute blade
  Interventions: Device: Alcon 25Gauge, 5,000 cuts per minute Ultravit cutter

INTERVENTIONS:
Device: Alcon 25Gauge, 10,000 cuts per minute Ultravit cutter — a proprietary Vitrector from Alcon for the use on the Constellation system
  Arms: 10k 25G cutter
Device: Alcon 25Gauge, 5,000 cuts per minute Ultravit cutter — a proprietary Vitrector from Alcon for the use on the Constellation system
  Arms: 5k 25G cutter

SUMMARY:
As technology advances, vitrectomy cutters are smaller and cut rates have become faster. In this prospective study, the vitrectomy efficiency and safety between 5,000 cuts per minute with 10,000 cuts per minute are compared

DETAILED DESCRIPTION:
Purpose:

This study aims to compare the performance of the Alcon 25+® UltraVit® 5000 cpm vitrectomy probe versus the 25+® Ultravit 10,000 cpm® beveled tip, dual drive vitrectomy probe. The safety profile and efficiency were compared.

Method:

Prospective, randomised study. Consecutive patients from January 2019 to August 2019 requiring vitrectomy for retinal detachment, epiretinal membrane, vitreous haemorrhage, and macula hole were randomized into either the 10K or 5K vitrectomy group. Both groups underwent vitrectomy using the proportional vacuum mode with the cut rate set at the fastest rate. Patients with previous vitrectomy, other ocular diseases (glaucoma, corneal disease, or significant corneal opacities), or trauma were excluded from the study. The primary endpoint was vitrectomy time, while secondary endpoints included posterior vitreous detachment time, intraoperative complications, and number of instruments used. The preoperative, postoperative 1 month and 3 month best corrected visual acuity (BCVA), and complications were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients over the age of 18 requiring vitrectomy for vitreous haemorrhage (VH), epiretinal membrane (ERM), macular hole (MH), dislocated lens, rhegmatogenous retinal detachment and diabetic tractional retinal detachment were randomized into the study from January 2019 till August 2019

Exclusion Criteria:

* Patients with ocular comorbidities affecting surgical view including corneal opacities or scar, previous vitrectomy, history of trauma or requiring silicone oil were excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Vitrectomy time | 1 day
  The time needed to remove all vitreous

SECONDARY OUTCOMES:
Safety and complications | up to 6 months
  Associated Intraoperative and post operative complications
Number of instruments used | 1 Day
  The total number of additional instruments used (scissors, forceps, etc)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No